CLINICAL TRIAL: NCT02273700
Title: Evaluation of Plasma Modifications Associated With Rivaroxaban® Treatment for Stroke Prevention in Patients With Atrial Fibrillation
Brief Title: Plasma Modifications Associated With Rivaroxaban® Treatment for Stroke Prevention
Acronym: Naco_Nîmes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2014/GL-01; 2014-A00516-41 (Other: RCB number)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
Keywords: Xarelto®; protein/peptide profiles
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- the Study Population: The study population consists of patients in the cardiology department at the Nîmes University Hospital with non-valvular atrial fibrillation and who are candidates for treatment with a direct oral anticoagulant: Rivaroxaban (Xarelto®). Patients will be selected according to criteria designed to result in a homogeneous population (associated anticoagulants, etc., see below). For this study, patients must not have had a direct oral anti-Xa (activated Factor 10) in the 6 months preceding enrollment.
  Intervention: Rivaroxaban
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Patients are observed during their first month of Rivaroxaban (Xarelto®) treatment, which is part of their routine care.
  Other Names: (Xarelto®)

SUMMARY:
The main objective of this pilot study is to investigate the protein / peptide plasma profiles before and after treatment with a direct anti-Xa (activated Factor 10) in patients with non-valvular atrial fibrillation to better understand the mechanisms of action of these molecules and perform exploratory analyses concerning proteins whose concentrations change after starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient was correctly informed about the study, its implementation, objectives, associated restrictions and patient rights
* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 1 month of follow-up
* The patient has non-valvular atrial fibrillation that was diagnosed within the last 3 months. Documentation of atrial fibrillation by a 12-lead ECG, an ECG rhythm strip, atrial fibrillation episode lasting at least 30 seconds.
* The patient has a CHA2-DS2-VASc score = 1, that is to say the presence of at least one of the following risk factors: (1) congestive heart failure or moderate to severe systolic dysfunction of the left ventricle; (2) history of systolic blood pressure> 160 mmHg; (3) diabetes; (4) history of ischemic stroke or systemic embolism; (5) vascular disease (myocardial infarction, arterial disease); (6) age > 65 years; (7) female.
* The patient will start Rivaroxaban (Xarelto®) at the Nîmes University Hospital

Exclusion Criteria:

* The patient is participating in another interventional study
* The patient has participated in another interventional study within the past three months
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Presence of a mechanical heart valve or valve disease
* Patient who recieved another new direct oral anticoagulant other than Xarelto® in the previous three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients in the cardiology department at the Nîmes University Hospital with non-valvular atrial fibrillation and who are candidates for treatment with a direct oral anticoagulant: Rivaroxaban (Xarelto®). Patients will be selected according to criteria designed to result in a homogeneous population (associated anticoagulants, etc., see below). For this study, patients must not have had a direct oral anti-Xa (activated Factor 10) in the 6 months preceding enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The percent change in plasma protein/peptide profiles after one month of treatment versus before treatment | 1 month (between days 28 to 35) versus baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Lavigne-Lissalde, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France